CLINICAL TRIAL: NCT06201988
Title: Assessing Patient Engagement and Understanding in Hepatic Encephalopathy Clinical Research
Brief Title: Revealing Engagement Patterns Among Hepatic Encephalopathy Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 67278255
Record Dates: First submitted 2023-12-29; First posted 2024-01-11 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Hepatic Encephalopathy
Keywords: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the influences behind patient choices regarding involvement, discontinuation, or re-engagement in hepatic encephalopathy clinical trials. Uncovering these factors is essential to enhance the relevance and efficacy of future research endeavors.

In essence, this trial aims to deepen understanding of the factors influencing participation in hepatic encephalopathy clinical trials. Elevating participation rates could expedite the development of innovative treatments for this challenging condition.

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent
* Aged ≥ 18 years old
* No prior treatment for hepatic encephalopathy

Exclusion Criteria:

* Participant is actively receiving study therapy in another
* Inability to provide written informed consent
* Women of childbearing potential without a negative pregnancy test; or women who are lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatic encephalopathy who are actively considering enrolling in a clinical study, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to join in a hepatic encephalopathy clinical trial | 3 months
Number of hepatic encephalopathy patients who remain in clinical trial until completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nardelli S, Gioia S, Faccioli J, Riggio O, Ridola L. Hepatic encephalopathy - recent advances in treatment and diagnosis. Expert Rev Gastroenterol Hepatol. 2023 Mar;17(3):225-235. doi: 10.1080/17474124.2023.2183386. Epub 2023 Feb 26. PMID 36843291
- [Background] Gairing SJ, Mangini C, Zarantonello L, Gioia S, Nielsen EJ, Danneberg S, Gabriel M, Ehrenbauer AF, Bloom PP, Ripoll C, Sultanik P, Galle PR, Labenz J, Thabut D, Zipprich A, Lok AS, Weissenborn K, Marquardt JU, Lauridsen MM, Nardelli S, Montagnese S, Labenz C. Prevalence of Minimal Hepatic Encephalopathy in Patients With Liver Cirrhosis: A Multicenter Study. Am J Gastroenterol. 2023 Dec 1;118(12):2191-2200. doi: 10.14309/ajg.0000000000002251. Epub 2023 Mar 20. PMID 36940426
- [Background] Bureau C, Thabut D, Jezequel C, Archambeaud I, D'Alteroche L, Dharancy S, Borentain P, Oberti F, Plessier A, De Ledinghen V, Ganne-Carrie N, Carbonell N, Rousseau V, Sommet A, Peron JM, Vinel JP. The Use of Rifaximin in the Prevention of Overt Hepatic Encephalopathy After Transjugular Intrahepatic Portosystemic Shunt : A Randomized Controlled Trial. Ann Intern Med. 2021 May;174(5):633-640. doi: 10.7326/M20-0202. Epub 2021 Feb 2. PMID 33524293

DOCUMENTS (1):
  • Informed Consent Form (2023-12-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT06201988/ICF_000.pdf